CLINICAL TRIAL: NCT04982705
Title: A Placebo- and Active-controlled, Randomised, Double-blind, Dose-escalation Phase I Study of IDG-16177 for the Evaluation of Its Safety and Pharmacokinetics With the Exploration on Its Pharmacodynamics and Efficacy
Brief Title: IDG-16177 for the Evaluation of Its Safety and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDG16177-T2DM-101; 2021-001082-21 (EudraCT Number)
Record Dates: First submitted 2021-07-05; First posted 2021-07-29 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes
Keywords: T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- [Part 1.1] IDG-16177 (Experimental): 6 subjects in each cohort (Cohort 1-5). The SAD study (Part 1.1) will consist of 5 cohorts of 8 healthy subjects who will be randomised to receive a single oral dose of IDG-16177 or placebo (6 active treatments and 2 placebo/3:1 ratio). Subjects in Cohort 4 will participate in a food-effect study.
  Interventions: Drug: [Part 1.1] IDG-16177
- [Part 1.1] Placebo of IDG-16177 (Placebo Comparator): 2 subjects in each cohort (Cohort 1-5). The SAD study (Part 1.1) will consist of 5 cohorts of 8 healthy subjects who will be randomised to receive a single oral dose of IDG-16177 or placebo (6 active treatments and 2 placebo/3:1 ratio). Subjects in Cohort 4 will participate in a food-effect study.
  Interventions: Drug: [Part 1.1] Placebo of IDG-16177
- [Part 1.2] IDG-16177 (Experimental): 8 subjects in each cohort (Cohort 6-8). The MAD study (Part 1.2) will consist of 3 cohorts of 10 healthy subjects (8 active treatments and 2 placebo/4:1 ratio), each receiving an oral dose of IDG-16177 or placebo.
  Interventions: Drug: [Part1.2] IDG-16177
- [Part 1.2] Placebo (Placebo Comparator): 2 subjects in each cohort (Cohort 6-8). The MAD study (Part 1.2) will consist of 3 cohorts of 10 healthy subjects (8 active treatments and 2 placebo/4:1 ratio), each receiving an oral dose of IDG-16177 or placebo (QD).
  Interventions: Drug: [Part 1.2] Placebo of IDG-16177
- [Part 2] IDG-16177 (Experimental): This part will consist of 3 separate arms of 8 patients per arm. Each arm will receive one of the following treatments: IDG-16177, placebo or DPP-4i as comparator.
  Interventions: Drug: [Part 2] IDG-16177
- [Part 2] Placebo (Placebo Comparator): This part will consist of 3 separate arms of 8 patients per arm. Each arm will receive one of the following treatments: IDG-16177, placebo or DPP-4i as comparator.
  Interventions: Drug: [Part 2] Placebo of IDG-16177
- [Part 2] Sitagliptin (Active Comparator): This part will consist of 3 separate arms of 8 patients per arm. Each arm will receive one of the following treatments: IDG-16177, placebo or DPP-4i as comparator (1:1:1 ratio).
  Interventions: Drug: [Part 2] Sitagliptin

INTERVENTIONS:
Drug: [Part 1.1] IDG-16177 — [Part 1.1] Subjects will receive a single oral dose of IMP. Dose strenght for each cohort (Cohort 1-5) is planned as 0.5, 1, 2, 5, 10mg, respectively.
  Arms: [Part 1.1] IDG-16177
Drug: [Part 1.1] Placebo of IDG-16177 — [Part 1.1] subjects will receive a single oral dose of IMP.
  Arms: [Part 1.1] Placebo of IDG-16177
Drug: [Part 2] Sitagliptin — Administration of Sitagliptin 100mg once daily for 4 weeks.
  Arms: [Part 2] Sitagliptin
Drug: [Part1.2] IDG-16177 — [Part 1.2] Administration once daily for 14 days; Dose strenght for each cohort (Cohort 6-8) is planned as ≤ 2, ≤ 4, ≤ 8mg, respectively.
  Arms: [Part 1.2] IDG-16177
Drug: [Part 2] IDG-16177 — [Part 2] Administration once daily for 4 weeks.
  Arms: [Part 2] IDG-16177
Drug: [Part 1.2] Placebo of IDG-16177 — [Part 1.2] Administration once daily for 14 days.
  Arms: [Part 1.2] Placebo
Drug: [Part 2] Placebo of IDG-16177 — [Part 2] Administration once daily for 4 weeks.
  Arms: [Part 2] Placebo

SUMMARY:
This is a Phase I, first-in-human, randomised, double-blinded, placebo-and active-controlled study to assess the safety, tolerability, PK, PD, efficacy, and food-effect of IDG-16177 in healthy male subjects and patients with T2DM at different dose levels.

DETAILED DESCRIPTION:
This study consists of 2 parts: Part 1 is a dose-escalation study in healthy male subjects in single ascending dose (SAD) (Part 1.1) including food-effect and multiple ascending dose (MAD) (Part 1.2) cohorts to determine the highest allowable dose (HAD) for patients with T2DM; and Part 2 is a placebo- and active-controlled efficacy exploration in patients with T2DM, insufficiently controlled with metformin alone.

ELIGIBILITY:
Inclusion Criteria:

[Part 1 and Part 2] Subjects/Patients who meet the following criteria will be considered eligible to participate in Part 1 or Part 2 of the clinical study:

1. Subject voluntarily/Patient agrees to participate in this study and signs an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent prior to performing any of the Screening Visit procedures. 2. Subject/Patient is able to understand the nature of the clinical study. 3. Subject/Patient is able to read and speak German. 4. Subject/Patient is able to communicate satisfactorily with the Investigator and study team and follow the entire requirements of the clinical study. [Part 1] Subjects who meet the following criteria will be considered eligible to participate in Part 1 of the clinical study:

1. Healthy male subjects aged 19 to 55 years at the time of Screening.
2. Subject weighs at least 60 kg and has a body mass index (BMI)between 18.5 and 29.9 kg/m2, inclusive, at Screening.
3. Subject who is healthy and judged to be eligible to participate in the study at the Screening test (based on medical history, physical examination, vital sign, 12 lead ECG, and laboratory test including serology test).

[Part 2] Patients who meet the following criteria will be considered eligible to participate in Part 2 of the clinical study:

1. Male patients aged 18 to 70 years at the time of Screening.
2. Patient with T2DM who is taking metformin monotherapy as their only anti hyperglycemic treatment. Metformin dose must be stable, defined as no change in the treatment, including dose, for at least 2 months prior to the screening visit.
3. Has a HbA1c level at Screening between 7.5% and 10.0%.
4. Has a fasting plasma glucose level less than 13.3 mmol/L at Screening.
5. Has a fasting C-peptide concentration greater than or equal to 0.8 ng/mL at Screening.
6. If patient takes any chronic medications, the dose of these medications must have been stable (no change in dose or drug) for at least 4 weeks prior to Screening.
7. Is able and willing to monitor glucose with a home glucose monitor and consistently record his blood glucose concentrations.
8. Patient weighs at least 60 kg and has a BMI between 18.5 and 35 kg/m2, inclusive, at Screening.

Exclusion Criteria:

[Part 1 and Part 2] Subjects/Patients who meet one or more of the following criteria will not be considered eligible to participate in Part 1 or Part 2 of the clinical study:

1. Subject/Patient is an employee or a family member of the Sponsor or the involved CRO.
2. Vulnerable subject (i.e., persons under any administrative or legal supervision or persons kept in detention).
3. Subject/Patient who has a positive reverse transcription polymerase chain reaction (RT PCR) test for SARS-CoV-2 prior to randomisation.
4. Subject/Patient who has clinical signs and symptoms consistent with SARS-CoV-2 infection; eg, fever, dry cough, dyspnea, sore throat, fatigue, or positive SARS-CoV-2 test result within 2 weeks prior to Screening.
5. Subject/patient who had a severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated).
6. Recent (within previous 14 days) exposure to someone who has COVID-19 symptoms or positive test result.
7. Subject who has currently acute disease with active symptoms.
8. History of clinically significant hypersensitivity reaction to any drugs or additives.
9. Subjects who have a history of any gastrointestinal disease (Crohn's disease, ulcerative colitis, acute or chronic pancreatitis) or gastrointestinal surgery (excluding simple appendectomy or herniotomy) which can affect the absorption of drugs.
10. Subject who has participated in a clinical trial or bioequivalence test and have been administered in a product within 60 days or within 5 halflives of the drug, whichever is longer before the first study drug administration.
11. Subject who have taken inducer or suppressor of metabolic enzymes such as barbiturates in 30 days before the first study drug administration.
12. Subject who have donated whole blood in 60 days or who have donated plasma in 20 days before the first study drug administration.
13. Subjects who have had any prescribed medicine or herbal medicine or who have had non-prescription medicine or vitamins within 7 days or 5 half lives before the first study drug administration, whichever is longer, except for occasional intake of paracetamol. Subjects who have received a SARS-CoV-2 vaccination within 4 weeks prior to screening or plan to be vaccinated during the study.
14. Has a history of drug abuse or a history of alcohol abuse within 2 years prior to Screening.
15. Subject who do not agree to be sexually abstinent or to use a condom with spermicide when engaging in sexual activity and to not donate sperm from the first administration of study drug, during the study, and for 14 days following completion of the study (Section 5.4.4).
16. Subject who is judged to be not eligible by the Investigator for any other reason.
17. Has a positive test result for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV).
18. Has a total bilirubin > 1.5 × ULN at Screening.
19. Has abnormal thyroid-stimulating hormone levels. [Part 1] Subjects who meet one or more of the following criteria will not be considered eligible to participate in Part 1 of the clinical study:
20. Subject who has abnormal vital signs, confirmed by repeat measurement at screening:

    * systolic blood pressure (SBP) outside 90 - 139 mmHg
    * diastolic blood pressure (DBP) outside 50 - 89 mmHg
    * pulse rate outside 50 - 90 bpm.
21. Abnormal 12-lead ECG, confirmed by repeat measurement, unless considered not clinically significant by Investigator. QTcF > 450 ms, QRS ≥ 120 ms, PR > 220 ms at Screening.
22. Has an estimating glomerular filtration rate (eGFR) less than or equal to 80 mL/min using the chronic kidney disease epidemiology collaboration (CKD EPI) at Screening.
23. History of clinically significant gastrointestinal, renal, hepatic, neurologic, haematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, musculoskeletal, or cardiovascular disease or any other condition. [Part 2] Patients who meet one or more of the following criteria will not be considered eligible to participate in Part 2 of clinical study:
24. Has systolic blood pressure (BP) greater than 160 mm Hg or diastolic pressure greater than 100 mm Hg at Screening or baseline, confirmed by repeat measurement.
25. Has history of cancer. A history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed.
26. Has a creatine phosphokinase level ≥ 5 × upper limit of normal (ULN) at Screening.
27. Has alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≥ 2 × ULN at Screening, confirmed by repeat measurement.
28. Has a haemoglobin level ≤ lower limit normal (LLN) for men of the local laboratory at Screening, confirmed by repeat measurement.
29. The subject has a serum triglyceride level ≥ 1.5 × ULN at Screening.
30. Has an eGFR less than or equal to 60 mL/min using the CKD EPI at Screening.

Ages: 19 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-11-09 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
AEs/serious AEs (SAEs) | Throughout study duration, up to 9 weeks
  Incidence and severity of adverse event
Percentage of subjects with clinically significant change from baseline in vital signs | Throughout study duration, up to 9 weeks
Percentage of subjects with clinically significant change from baseline in electrocardiogram (ECG) | Throughout study duration, up to 9 weeks
Percentage of subejcts with clinically significant change from baseline in safety laboratory test results | Throughout study duration, up to 9 weeks

SECONDARY OUTCOMES:
Maximum concentration of IDG-16177(Cmax) | Throughout study duration, up to 9 weeks
Time of maximum plasma IDG-16177 concentration (Tmax) | Throughout study duration, up to 9 weeks
Area under the concentration-time curve (AUC) | Throughout study duration, up to 9 weeks
Terminal elimination rate constant (λz) | Throughout study duration, up to 9 weeks
Terminal elimination half-life calculated as: ln2/λz (T½) | Throughout study duration, up to 9 weeks
Apparent total clearance of the drug from plasma after oral administration (CL/F) | Throughout study duration, up to 9 weeks
Cumulative urinary excretion from time 0 to time t (Ae0-t) | Throughout study duration, up to 9 weeks
Renal clearance of the drug from plasma (CLR) | Throughout study duration, up to 9 weeks
Accumulation ratio (Rac) | Throughout study duration, up to 9 weeks
Apparent volume of distribution following oral administration (Vd/F) | Throughout study duration, up to 9 weeks

OTHER OUTCOMES:
Insulin | Through the treatment; Plasma concentration will be observed at baseline and 0.25, 0.5, 1, 1.5, 2, 3 and 4 hours after dose
  plasma concentration
proinsulin | Through the treatment; Plasma concentration will be observed at baseline and 0.25, 0.5, 1, 1.5, 2, 3 and 4 hours after dose
  plasma concentration
C-peptide | Through the treatment; Plasma concentration will be observed at baseline and 0.25, 0.5, 1, 1.5, 2, 3 and 4 hours after dose
  plasma concentration
Glucagon | Through the treatment; Plasma concentration will be observed at baseline and 0.25, 0.5, 1, 1.5, 2, 3 and 4 hours after dose
  plasma concentration
Glucose | Through the treatment; Plasma concentration will be observed at baseline and 0.25, 0.5, 1, 1.5, 2, 3 and 4 hours after dose
  plasma concentration
HbA1c level | Through the treatment; Days 8, 15 and 28
  Change from baseline in HbA1c level

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International GmbH Early Phase Clinical Unit Klinikum Westend, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided